CLINICAL TRIAL: NCT00000450
Title: Nalmefene Maintenance Treatment of Alcoholism
Brief Title: Naltrexone Maintenance Treatment of Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, Principal Investigator, The Scripps Research Institute
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAMAS10518; R01AA010518 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Naltrexone 50 mg was provided for 3 months to all study participants, who were masked regarding the identity of study medication. At 3 months, full and partial responders were randomized to an additional 9 months of double blind treatment with naltrexone or matched placebo. Full responders were defined as complete abstinence for the last six weeks of the acute phase. Partial responders were defined as having no more than 2 heavy drinking days in any given week and/or a 50% reduction in weekly alcohol consumption from baseline over the last six weeks of the acute phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Naltrexone and placebo were identical in appearance and packaging to preserve the double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naltrexone Tablet (Active Comparator)
  Interventions: Drug: Naltrexone Tablet
- Matched Placebo Tablet (Placebo Comparator)
  Interventions: Drug: Matched Placebo Tablet

INTERVENTIONS:
Drug: Naltrexone Tablet
  Other Names: Revia
  Arms: Naltrexone Tablet
Drug: Matched Placebo Tablet
  Other Names: Placebo
  Arms: Matched Placebo Tablet

SUMMARY:
The purpose of this study is to determine the long-term effectiveness of naltrexone treatment in alcohol-dependent patients who respond to short-term treatment. Those who respond to short-term treatment will be randomized to a 1-year, double-blind, placebo-controlled maintenance phase with a 6-month posttreatment followup.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence.
* Expresses a desire to cut down or stop drinking.

Exclusion Criteria:

* Currently meets criteria for dependence on substances other than alcohol.
* History of opiate dependence or evidence of current opiate use.
* Significant medical disorders that will increase potential risk or interfere with study participation.
* Liver function tests more than 3 times normal or elevated bilirubin.
* Female patients who are pregnant, nursing, or not using a reliable method of birth control.
* Inability to understand and provide a consent form.
* Treatment with an investigational drug during the previous month.
* Prior treatment with naltrexone.
* Chronic treatment with any narcotic-containing medications during the previous month.
* Sensitivity to naltrexone as evidenced by adverse drug experiences especially with narcotic containing analgesics or opioid antagonists.
* Current treatment with disulfiram.
* More than 6 weeks of abstinence.
* Meets criteria for a major psychiatric disorder and is in need of, or currently undergoing pharmacotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 1997-04-10 (Actual); Primary Completion 2002-02-13 (Actual); Study Completion 2002-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- Department of Psychiatry, University of Miami School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No